CLINICAL TRIAL: NCT06266559
Title: Efficacy Evaluation of Chang Geng Healthy Drink on Patients With Non-alcoholic Fatty Liver Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tse-Hung Huang, Principal Investigator, Clinical Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202101896A3
Record Dates: First submitted 2024-02-07; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Traditional Chinese Medicine; Brief Fatigue Inventory - Taiwanese Form; FibroScan
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial Drink Group (Experimental): Consume one bottle of Chang Geng Healthy Drink per day for the first eight weeks of the trial.
  Interventions: Other: Chang Geng Healthy Drink
- Subsequent Drink Group (Experimental): Consume one bottle of Chang Geng Healthy Drink per day for the last eight weeks of the trial.
  Interventions: Other: Chang Geng Healthy Drink

INTERVENTIONS:
Other: Chang Geng Healthy Drink — Chang Geng Healthy Drink consists of Zingiberis Rhizoma, Codonopsis pilosula, Atractylodis Macrocephalae Rhizoma, Poria cocos, Citri reticulatae Pericarpium

SUMMARY:
For non-alcoholic fatty liver disease, there is currently no effective treatment options. Traditional Chinese medicine (TCM) has a long history of treating liver diseases. However, TCM treatment methods are diverse, and there is currently a lack of high-quality clinical research to confirm the efficacy of Chinese herbal medicine. Thereafter, Chang-Gung Healthy Drink which is a TCM based healthy drink may be used to alleviate the clinical adverse event of non-alcoholic fatty liver disease patients.

DETAILED DESCRIPTION:
For non-alcoholic fatty liver disease, there is currently no effective treatment method. Some studies suggest that a low-calorie diet, exercise, weight loss, etc., may help alleviate clinical symptoms, but the evidence is inconsistent. Traditional Chinese medicine (TCM) has a long history of treating liver diseases, and the formation of non-alcoholic fatty liver disease may be due to liver depression and blood stasis caused by spleen-stomach disharmony. In treatment, traditional Chinese medicine usually focuses on soothing the liver, promoting qi circulation, activating blood circulation, and resolving blood stasis. However, TCM treatment methods are diverse, and there is currently a lack of high-quality clinical research to confirm the efficacy of Chinese herbal medicine. Thereafter, Chang-Gung Healthy Drink which is a TCM based healthy drink may be used to alleviate the clinical adverse event of non-alcoholic fatty liver disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged between 20 and 75 years old.
* Capable of understanding and signing the Informed Consent Form (ICF) document.
* Diagnosed by a physician with non-alcoholic moderate fatty liver.
* Liver function index, AST or ALT, elevated to 2 to 5 times the normal value for more than 1 month.

Exclusion Criteria:

* Diagnosed with alcoholic fatty liver, viral hepatitis, autoimmune hepatitis, Wilson's Disease, drug-induced hepatitis, or hemochromatosis.
* Currently suffering from major illnesses such as cancer, stroke, end-stage kidney disease, cirrhosis.
* Men who consume more than 140g of alcohol per week, or women who consume more than 70g of alcohol per week.
* Consuming other chinese herbal medicine.
* Pregnant or lactating women.
* Patients using lipid-lowering and diabetes medications.
* Patients with Covid-19.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-03-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue Visual Analogue Scale - Current fatigue level | 18 weeks
  Brief Fatigue Inventory - Taiwanese Form (BFI-T) with a scale from 0 (least fatigue) to 10 (most fatigue) assessing current fatigue level.
Fatigue Visual Analogue Scale - Other daily specific task fatigue level | 18 weeks
  Brief Fatigue Inventory - Taiwanese Form (BFI-T) with a scale from 0 (least fatigue) to 10 (most fatigue) assessing other daily specific task fatigue level.
Laboratory Data (Linver Function Index) | 18 weeks
  Aspartate Aminotransferase, Alanine transaminase
Liver stiffness measurement (kPa) | 18 weeks
  FibroScan - A Non-invasive Liver Fibrosis Assessment Device. Assess liver stiffness level (F1 - F4) with liver stiffness measurement (LSM) score.
Controlled attenuation parameter (dB/m) | 18 weeks
  FibroScan - A Non-invasive Liver Fibrosis Assessment Device. Assess Liver steatosis level (S0 - S3) according to controlled attenuation parameter (CAP) score

SECONDARY OUTCOMES:
Number of Participants With Clinical Significant Adverse Avent (Safety Measures) | 18 weeks
  Number of participants with significant adverse event during the trial. Also record the category and severity grade of adverse event according to CTCAE Version 5.0